CLINICAL TRIAL: NCT00294892
Title: The Effect of Single Dose Carbamazepine on the Pharmacokinetics of Single Dose Nevirapine (Viramune, NVP) and Development of NVP Resistance, PMTCT Program of Moshi, Tanzania (VITA1)
Brief Title: Pharmacokinetics Study on Nevirapine Resistance in Tanzania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITA1
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections
Keywords: HIV; mother to child transmission; MTCT; nevirapine resistance; pharmacokinetics; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Carbamazepine; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbamazepine (Active Comparator): An oral dose of 400mg Carbamazepine is added to the 200mg oral dose Nevirapine intake prior delivery
  Interventions: Drug: carbamazepine and nevirapine
- Nevirapine (Placebo Comparator): Standard therapy of 200mg Nevirapine oral prior to delivery
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: carbamazepine and nevirapine — Carbamazepine 400mg and Nevirapine 200mg are taken just before delivery during labor.
  Arms: Carbamazepine
Drug: Nevirapine — Nevirapine 200mg is taken prior to delivery during labor.
  Arms: Nevirapine

SUMMARY:
Primary

* pharmacokinetics of single dose nevirapine
* the effect of single dose carbamazepine on the pk of single dose nevirapine
* resistance against nevirapine before and after.
* follow-up on HIV status newborns
* relation between nevirapine levels in cord blood and plasma

Secondary

* safety of single dose nevirapine and nevirapine/carbamazepine

Hypothesis:

Single dose carbamazepine decreases development of resistance to nevirapine in HIV positive pregnant Tanzanian women by decreasing nevirapine half-life.

DETAILED DESCRIPTION:
Without the use of preventative measures, the risk of mother-to-child transmission (MTCT) of HIV-1 is estimated to vary between 25 and 48%. The regimen of single dose of nevirapine to the mother just before delivery and a single dose of nevirapine to the newborn within 24 - 72 hours after birth reduces the risk of MTCT by 50%, is affordable in many situations and is therefore standard of care in many African countries, like Tanzania. Recent studies, however, have shown that this single dose to the mother can induce the occurrence of nevirapine resistance in a large number of mothers. The mechanism of occurrence of nevirapine resistance already after a single dose is most likely related to the long elimination half-life of the drug. The subtherapeutic plasma levels present the perfect environment for the occurrence of resistance as the concentrations are subinhibitory for several days.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* antiretroviral naive
* not intending to relocate out of area during study
* willing to adhere to follow up scheme
* ability and willing to give written consent
* pregnant between 18 and 40 years
* willing and able to regularly attend the Antenatal clinic

Exclusion Criteria:

* serious illness that requires systemic treatment or hospitalization
* any condition that would compromise subject's ability to participate
* previously treated for HIV with antiretroviral agents, including single dose nevirapine used for MTCT
* inability to understand the nature and extent of the trial and procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2006-02; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Cord blood will be taken less than 30 minutes after delivery | 0 - 30 min after delivery
Blood samples from mother will be taken less than 30 minutes after delivery to measure viral load and CD4 count. | 0 - 30 min after delivery
Blood samples will be drawn from mother and child at week 1 (day 6-8), week 2 (day 13-15) and week 3 (day 20-22) | day 6 - 22 after delivery
From all samples plasma nevirapine and if applicable carbamazepine levels will be determined in women and newborns. | 0 30 min after delivery - week 3 after delivery

CONTACTS AND LOCATIONS:
Overall Officials: David M. Burger, Dr., Principal Investigator — Radboud University (RUNMC)
Locations (1):
- Kilimanjaro Christian Medical College, Moshi, Tanzania

REFERENCES:
- [Derived] Muro EP, Fillekes Q, Kisanga ER, L'homme R, Aitken SC, Mariki G, Van der Ven AJ, Dolmans W, Schuurman R, Walker AS, Gibb DM, Burger DM. Intrapartum single-dose carbamazepine reduces nevirapine levels faster and may decrease resistance after a single dose of nevirapine for perinatal HIV prevention. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):266-73. doi: 10.1097/QAI.0b013e31824234d8. PMID 22134145
- See also: J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):266-73. Intrapartum single-dose carbamazepine reduces nevirapine levels faster and may decrease resistance after a single dose of nevirapine for perinatal HIV prevention. — http://journals.lww.com/jaids/Abstract/2012/03010/Intrapartum_Single_Dose_Carbamazepine_Reduces.7.aspx